CLINICAL TRIAL: NCT00691951
Title: Comparative Effects of Budesonide and Budesonide/Formoterol (Symbicort) on Asthma Control in Smoking Asthmatic Subjects: A Pilot Study
Brief Title: Effects of Budesonide & Budesonide/Formoterol on Smoking Asthmatic Subjects
Acronym: D5890L00013
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Louis-Philippe Boulet, Laval University
Other Study IDs: Symbicort smokers AZ
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate

INTERVENTIONS:
Drug: budesonide and budesonide/formoterol

SUMMARY:
A reduced response to inhaled corticosteroids (ICS) has been reported in smoking compared to non-smoking asthmatic patients. However, the comparative response to other currently prescribed medications such as combination therapy of long-acting beta agonists and ICS remain to be further evaluated.

No significant differences were found between our group of subjects in regard to changes in asthma control pulmonary function and airway inflammation following budesonide or the association of budesonide with formoterol for a period of 2 months. This should be further explored in larger groups of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic non-smokers or ex-smokers (less than 10 pack/years)
* Asthmatic smokers (more than 5 cigarettes a day and more than 5 pack/years
* FEV1 greater than 70%
* No more than 3 doses of rescue medication (bronchodilator) per day

Exclusion Criteria:

* Mentally or legally incapacitated thus preventing informed consent from being obtained
* Other pulmonary disorder
* History of upper respiratory tract infection in the last month
* Pregnant or lactating women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Comparative changes before and after treatments in each group for Asthma Control Questionnaire (ACQ)

SECONDARY OUTCOMES:
Other control scores (ACSS score) and rescue B2 agonist need
Comparative changes in FEV1
Quality of life questionnaire
Morning and evening PEF
Total and differential cell counts in induced sputum and ECP and MPO

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Hôpital du Sacré-Coeur de Montreal, Montreal, Quebec
  - Laval Hospital, Québec, Quebec